CLINICAL TRIAL: NCT03214042
Title: Efficacy and Safety of K-rod Dynamic Stabilization System in the Repair of Lumbar Degenerative Diseases: Study Protocol for a Prospective, Self-controlled, Clinical Trial
Brief Title: Efficacy and Safety of K-rod Dynamic Stabilization System in the Repair of Lumbar Degenerative Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shenyang Orthopedic Hospital (Other)
Responsible Party: Principal Investigator, Shuyi Gong, Principal Investigator, Shenyang Orthopedic Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShenyangOrthoH-01
Record Dates: First submitted 2017-07-09; First posted 2017-07-11 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Intervertebral Disk Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- trial group (Experimental): Sixty-seven patients with lumbar degenerative diseases were treated with K-rod dynamic stabilization system. All patients were followed for 2 years.
  Interventions: Device: K-rod dynamic stabilization system

INTERVENTIONS:
Device: K-rod dynamic stabilization system — Sixty-seven patients with lumbar degenerative diseases were treated with K-rod dynamic stabilization system. All patients were followed for 2 years. K-rod dynamic stabilization system was purchased from Biotech, USA, consisting of titanium alloy pedicle screw, titanium alloy line and polyether ether ketone (PEEK) shell between pedicle screw heads.

SUMMARY:
To conduct a prospective, single-center, self-controlled, clinical trial to verify the efficacy and safety of K-Rod dynamic stability system in the repair of lumbar degenerative diseases following 2 years follow-up, aiming to provide references for clinical treatment of lumbar degenerative diseases.

DETAILED DESCRIPTION:
Posterior internal fixation and fusion systems are still one of the main methods for the treatment of chronic back pain due to intervertebral disc degeneration, but adverse reactions, such as accelerated regression of adjacent segments, are often inevitable during the treatment.

At present, various pedicle screw-based posterior dynamic stability systems of the lumbar spine have become an alternative fusion therapy for lumbar degenerative diseases. Dynamic stability is defined to reduce the loading on the intervertebral disc/articular surfaces, to maintain movement under mechanical load, to limit the abnormal movement of the spinal segment, and to reduce the stress on the bone-screw interface dynamically and stably. An ideal fixation system will be stable enough to maximize the fusion rate without the need for excessive rigidity, as well as to maintain maximum load and physiological posture of the vertebral segment, thereby reducing the horizontal stress of the adjacent segment.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative lumbar spondylolisthesis (degree I)
* Nerve root canal or central spinal canal stenosis
* Accompanying nerve root pain and/or chronic back pain
* 32-76 years old
* Regardless of gender
* All patients or family members signed the informed consent

Exclusion Criteria:

* Systemic infection;
* Poor compliance and inability to complete the trial

Ages: 32 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Oswestry dysfunction index scores | at month 24 after surgery
  To quantify disability for pain. The Oswestry Disability Index questionnaire contains ten questions concerning intensity of pain, ability to take care of oneself, lifting, ability to walk, ability to sit, ability to stand, sleep quality, sexual life, social life, and ability to travel. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability.

SECONDARY OUTCOMES:
Lumbar lordosis angle | at month 24 after surgery
  The lumbar lordosis angle refers to an angle between the lower end plate of L1 and the upper end plate of S1 on the lateral X-ray.

CONTACTS AND LOCATIONS:
Overall Officials: Shuyi Gong, Principal Investigator — Shenyang Orthopedic Hospital

IPD SHARING:
Plan to Share IPD: Undecided